CLINICAL TRIAL: NCT01004497
Title: A Phase 2 Multicenter Study of First-line Dasatinib Plus Conventional Chemotherapy in Adults With Newly Diagnosed Philadelphia Chromosome-Positive Acute Lymphoblastic Leukemia
Brief Title: First-line Dasatinib Plus Conventional Chemotherapy in Adults With Newly Diagnosed Ph-Positive ALL
Acronym: ALL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Seok Lee, Professor, The Catholic University of Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KC09MIMS0255
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia, adult, dasatinib
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib; Cyclophosphamide; Vincristine; Daunorubicin; Dexamethasone; dexamethasone 21-phosphate; Cytarabine; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Modified Hyper-CVAD + Dasatinib (Experimental): Dasatinib: 100 mg once daily, PO, for 4 weeks Cyclophosphamide: 300 mg/m2, IV, every 12 hours, days 1~3 Vincristine: 1.4 mg/m2/day (maximum 2 mg/day), IV, days 4 & 11 Daunorubicin: 45 mg/m2/day, IV, days 4 & 11 Dexamethasone: 40 mg/day, IV, days 1~4 & days 11~14 Cytarabine: 2 g/m2, IV, every 12 hours, days 1~5 Mitoxantrone: 12 mg/m2/day, IV, days 1~2
  Interventions: Drug: Dasatinib; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Daunorubicin; Drug: Dexamethasone; Drug: Cytarabine; Drug: Mitoxantrone

INTERVENTIONS:
Drug: Dasatinib — After the completion of each induction and consolidation chemotherapy with recovery of leukocyte and platelet counts, dasatinib will be given as an alternative manner: 100 mg by mouth once daily for 4 weeks
  Other Names: Sprycel
Drug: Cyclophosphamide — 300 mg/m2, IV for 2 hours, every 12 hours x 6 doses, days 1-3
  Other Names: Endoxan
Drug: Vincristine — 1.4 mg/m2/day (maximum 2 mg/day), IV for 30 minutes, days 4 & 11
  Other Names: Vincristine sulfate
Drug: Daunorubicin — 45 mg/m2/day, IV for 1 hour, days 4 & 11
  Other Names: Cerubidine
Drug: Dexamethasone — 40 mg/day, IV push, days 1-4 & days 11-14
  Other Names: Dexamethasone disodium phosphate
Drug: Cytarabine — 2 g/m2, IV for 3 hours, every 12 hours x 10 doses, days 1-5
  Other Names: Cytosar U
Drug: Mitoxantrone — 12 mg/m2/day, IV for 30 minutes, days 1-2
  Other Names: Mitrone

SUMMARY:
The main aim of the present study is to evaluate the clinical efficacy of first-line dasatinib plus conventional chemotherapy for newly diagnosed Ph-positive acute lymphoblastic leukemia. In this study, the investigators will analyze the clinical outcomes for entire patient population as well as those for transplants, respectively. In addition, the results of this study will be compared to those of the investigators current study (imatinib plus conventional chemotherapy). The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Recent clinical trials on imatinib in combination with cytotoxic agents as a front-line treatment, have demonstrated an improved complete remission (CR) rate and a better outcome in adults with Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph-positive ALL). Previously, we also demonstrated the positive impact of first-line imatinib interim therapy on the outcome of allogeneic stem cell transplantation (SCT) in adults with Ph-positive ALL. Nevertheless, a substantial proportion of patients continue to die as a result of disease progression. Recently, we demonstrated that a reduction in BCR-ABL transcript levels of at least 3 log after the completion of imatinib therapy was found to be the most powerful predictor of lower relapse and better disease-free survival after allogeneic SCT. In the light of disease aggressiveness and recurrence, mainly as a result of the outgrowth of leukemic subclones with imatinib-resistant BCR-ABL mutations, an improved strategy to induce more effective leukemic cell clearance during the pretransplantation treatment course is clearly needed.

Dasatinib, a potent dual BCR-ABL/SRC family kinase inhibitor, demonstrated 325-fold greater activity against native BCR-ABL compared with imatinib and has shown efficacy against all imatinib-resistant BCR-ABL mutations with the exception of T315I. According to the START-L (SRC/ABL Tyrosine Kinase Inhibition Activity: Research Trials of Dasatinib) trial, dasatinib (70 mg twice daily) induced rapid hematologic and cytogenetic responses in a substantial proportion of patients with imatinib-resistant or intolerant Ph-positive ALL (hematologic CR rate, 33%; major cytogenetic response rate, 57%; cytogenetic CR rate, 54%). However, the median duration of a major cytogenetic response was 6.9 months. Considering this kinetics of resistance, it is felt likely that dasatinib monotherapy is not sufficient as a first-line treatment for Ph-positive ALL.

Allogeneic SCT clearly benefits certain high-risk patients, such as those with Ph-positive ALL or those that show a poor initial response to chemotherapy, and long-term survival rates with SCT are markedly increased when patients are in CR. Recent studies suggest that among adults with ALL, transplantation from a matched unrelated donor could yield results similar to those achieved by matched related donor transplantation. While unrelated donor transplants are generally associated with more transplant-related complications than matched sibling transplants, a compensatory decrease in relapse rates due to a strong graft-versus-leukemia effect has narrowed the gap between the two approaches. In addition, reduced-intensity conditioning allogeneic SCT is increasingly being used for patients who are considered poor candidates for myeloablative conditioning SCT because of their advanced age or other concurrent medical conditions. Two recent reports of patients undergoing a transplant using related or unrelated donor and a reduced-intensity conditioning regimen (fludarabine plus melphalan) showed an optimistic outcome in a group of patients with ALL either at high risk during first CR or who were transplanted after achieving a subsequent CR. Recently, we also demonstrated an evidence of positive role of reduced-intensity conditioning SCT for the management of high-risk adult ALL who are ineligible for myeloablative transplantation with low leukemic cell burden (especially in first CR) through a prospective analysis (phase 2 study). From this point of view, the role of first-line dasatinib plus conventional chemotherapy followed by allogeneic SCT should be clarified in the era of targeted drugs.

Recently, the results of the phase 3 study in patients with chronic phase-chronic myeloid leukemia suggest that dasatinib (100 mg q.d.) offers the most favorable overall benefit-risk assessment. On the basis of these results, dasatinib will be administered orally at 100 mg once a day in this study.

Induction regimen: "Modified Hyper-CVAD"

* Cyclophosphamide 300 mg/m2, IV for 2 hours, every 12 hours x 6 doses, days 1-3
* Vincristine 1.4 mg/m2/day (maximum 2 mg/day), IV for 30 minutes, days 4 & 11
* Daunorubicin 45 mg/m2/day, IV for 1 hour, days 4 & 11
* Dexamethasone 40 mg/day, IV push, days 1~4 & days 11-14

First consolidation regimen: "Cytarabine and Mitoxantrone"

* Cytarabine 2 g/m2, IV for 3 hours, every 12 hours x 10 doses, days 1-5
* Mitoxantrone 12 mg/m2/day, IV for 30 minutes, days 1-2

Second consolidation regimen: "Modified Hyper-CVAD"

* Cyclophosphamide 300 mg/m2, IV over 2 hours, every 12 hours x 6 doses, days 1-3
* Vincristine 1.4 mg/m2/day (maximum 2 mg/day), IV for 30 minutes, days 4 & 11
* Daunorubicin 45 mg/m2/day, IV for 1 hour, days 4 & 11
* Dexamethasone 40 mg/day, IV push, days 1-4 & days 11-14

Dose of chemotherapeutic drugs (except vincristine, dexamethasone, and etoposide) will be reduced by 25% in patients aged between 50 and 59 years; and by 50% in patients 60 years or older. During the consolidation phase, serious toxicities (more than or equal to grade 3 non-hematologic toxicities) will require subsequent dose reductions of 25% to 50% at the attending physician's discretion.

Central nervous system prophylaxis will be performed by intrathecally administering triple agents (methotrexate 12 mg, cytarabine 40 mg, and hydrocortisone 50 mg; 6 times in total).

After the completion of each induction and consolidation chemotherapy with recovery of leukocyte and platelet counts, dasatinib will be given as an alternative manner (100 mg once daily by mouth for 4 weeks).

Dasatinib dose adjustment will be performed according to the guidelines for managing hematologic and nonhematologic adverse events during dasatinib treatment. Briefly,

1. Dose escalation will be permitted in patients with no hematologic CR (to 140 mg daily; 140 mg q.d. or 70 mg b.i.d.).
2. Dose reduction (to 80 mg daily; 80 mg q.d. or 40 mg b.i.d.) and interruption will be permitted after dasatinib-related grades 3-4 hematologic toxicity or grades 2-4 nonhematologic toxicity .

Dasatinib will be administered until disease progression or intolerable toxicity, as determined by the treating physician.

Patients with an HLA-matched or suitable donor will undergo allogeneic SCT.

Patients without a donor will undergo continuous consolidation (up to 4 courses) and maintenance therapy (dasatinib 100 mg once daily for up to 2 years as long as the patients remain in hematologic CR with stable MRD level).

The number of dasatinib plus conventional chemotherapy will be dependent on the speed of coordination process (for transplants) or the patient's tolerability (for non-transplants).

SCT from an HLA-matched sibling or a suitably matched (less than or equal to 2-allele mismatched) family or unrelated donor will be performed according to the policies of the participating institutions. A preparative regimen will be started 7 days after the last day of the dasatinib treatment.

No prophylactic dasatinib maintenance therapy is planned after SCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed acute lymphoblastic or biphenotypic leukemia (karyotypic or molecular evidence of Ph)
* Ages of 15-65 years
* Eastern Cooperative Oncology Group performance status of 0-2
* Adequate renal (serum creatinine less than 2 mg/dl, unless considered due to leukemia) and hepatic (serum bilirubin less than 3 mg/dl, unless considered due to leukemia) functions
* Adequate cardiac status (New York Heart Association Class less than or equal to 2)
* Signed informed consent

Exclusion Criteria:

* Pregnant and lactating women will not be eligible. Women of childbearing potential should have a negative pregnancy test prior to entering on the study.
* Active cardiac dysfunction (New York Heart Association Class more than or equal to 3), uncontrolled angina, myocardial infarction (within 6 months), congenital long QT syndrome, any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia or ventricular fibrillation), or prolonged QTc interval on pre-entry electrocardiogram (more than 470 msec)
* Patients with documented significant pleural or pericardial effusions unless they are thought to be secondary to their leukemia
* Patients with severe medical conditions that in the view of the investigator prohibits participation in the study
* Treatment with any other investigational antileukemic agents in the last 30 days before study entry

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-03; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine the clinical efficacy of dasatinib plus conventional chemotherapy for newly diagnosed Ph-positive ALL in terms of major molecular response rate | by the second 4-week dasatinib therapy

SECONDARY OUTCOMES:
To evaluate the long-term clinical outcomes (including transplant outcomes) in terms of treatment toxicity, relapse, disease-free survival, and overall survival | at 2 years after transplantation (for all transplants); at 2 years after starting dasatinib maintenance (for all non-transplants)

CONTACTS AND LOCATIONS:
Overall Officials: Seok Lee, M.D., Principal Investigator — Catholic BMT Center, Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (8):
- South Korea (8):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - St. Vincent's Hospital, The Catholic University of Korea, Suwon, Kyonggi-do
  - Yonsei University Severance Hospital, Seoul
  - Catholic BMT Center, Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Derived] Yoon JH, Yhim HY, Kwak JY, Ahn JS, Yang DH, Lee JJ, Kim SJ, Kim JS, Park SJ, Choi CW, Eom HS, Park SK, Choi SY, Kim SH, Kim DW, Lee S. Minimal residual disease-based effect and long-term outcome of first-line dasatinib combined with chemotherapy for adult Philadelphia chromosome-positive acute lymphoblastic leukemia. Ann Oncol. 2016 Jun;27(6):1081-1088. doi: 10.1093/annonc/mdw123. Epub 2016 Mar 6. PMID 26951627